CLINICAL TRIAL: NCT02034903
Title: Effect of Feed Warming Method on Feeding Tolerance in the Preterm Infant Born at Less Than 30 Weeks Gestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advocate Center for Pediatric Research (Other)
Collaborators: Wake Forest University Health Sciences (Other); Medela AG (Industry)
Responsible Party: Principal Investigator, Bonnie Satinover, RN-NIC, Clinician III, NICU, Advocate Center for Pediatric Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5283
Record Dates: First submitted 2014-01-08; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Enteral Feeding
Keywords: Enteral Feeding; Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard warming (No Intervention): Feeding warmed in water bath
- Commercial warmer (Experimental): Feedings warmed with a commercial warmer
  Interventions: Other: Feedings warmed with commercial warmer

INTERVENTIONS:
Other: Feedings warmed with commercial warmer
  Arms: Commercial warmer

SUMMARY:
The temperature of milk fed to infants in the Neonatal Intensive Care Unit (NICU) has been shown to vary greatly, and is influenced by individual provider practice. The clinical effect of varying milk temperatures on preterm infant feeding tolerance has not been well studied. The purpose of this study is to examine the effect of warming method, water bath versus commercial warmer and its impact on feeding tolerance. Sample population will include eighty-six infants born at 30-0/7 weeks or less, and admitted to the Neonatal Intensive Care Unit at Advocate Children's Hospital, Park Ridge within 48 hours of birth and remain in the study for a minimum of 28 days. After obtaining consent, eligible infants will be assigned to a control (water bath) or experimental (commercial warmer) group using a randomized sampling scheme. After warming, and just prior to feeding, milk temperatures will be taken and recorded by a trained data recorder. Feeding tolerance will be measured based on gastric residual volume and length of time required to achieve full feeds. Based upon the available evidence, the study investigators hypothesize that warming feeds to a consistent temperature range using commercially available milk warmer will improve feeding tolerance and decrease time to full feedings in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at less than or equal to 30 0/7 weeks gestation
* Infants will be enrolled within the first 48 hours of life

Exclusion Criteria:

* Gastrointestinal anomalies
* Lethal malformations
* Parental denial of consent or request for removal from study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Feeding intolerance | 168 completed feedings; approximately 28 days
  Feeding intolerance is defined by one or more of the following clinical observations:
  1. Abdominal distention defined as increase in abdominal girth > 1 cm. since previous nursing assessment
  2. Obvious blood in stool
  3. Persistent regurgitation (>3 consecutive feedings)
  4. Significant gastric residuals:
     1. 25-50% of feeding volume x 2 consecutive feeds
     2. > 50% of feeding volume x 1 feed

SECONDARY OUTCOMES:
Full enteral feeding | approximately 28 days
  The point in time that parenteral nutrition is discontinued based on the judgment that the infant's enteral intake is sufficient to continue growth and development.

CONTACTS AND LOCATIONS:
Locations (1):
- Advocate Children's Hospital, Park Ridge, Park Ridge, Illinois, United States